CLINICAL TRIAL: NCT07196774
Title: A Randomized, Open-label, Multicenter Phase III Study of SHR-A1811 Compared to Docetaxel+Carboplatin+Trastuzumab+Pertuzumab as a Neoadjuvant Therapy for the Initial Treatment of Early-stage or Locally Advanced HER2-positive Breast Cancer
Brief Title: A Trial of SHR-A1811 Compared to Other Antitumor Therapies as Neoadjuvant Treatments in Early-stage or Locally Advanced HER2-positive Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811-312
Record Dates: First submitted 2025-09-22; First posted 2025-09-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Early-stage or Locally Advanced HER2-positive Breast Cancer
MeSH Terms: interventions — Injections; Docetaxel; Trastuzumab; Carboplatin; pertuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-A1811 Group (Experimental)
  Interventions: Drug: SHR-A1811 for Injection
- Docetaxel+Carboplatin+Trastuzumab+Pertuzumab Group (Active Comparator)
  Interventions: Drug: Docetaxel injection; Drug: Trastuzumab Injection; Drug: Carboplatin for Injection; Drug: Pertuzumab Injection

INTERVENTIONS:
Drug: SHR-A1811 for Injection — SHR-A1811 for injection.
  Arms: SHR-A1811 Group
Drug: Docetaxel injection — Docetaxel injection.
  Arms: Docetaxel+Carboplatin+Trastuzumab+Pertuzumab Group
Drug: Trastuzumab Injection — Trastuzumab injection.
  Arms: Docetaxel+Carboplatin+Trastuzumab+Pertuzumab Group
Drug: Carboplatin for Injection — Carboplatin for injection.
  Arms: Docetaxel+Carboplatin+Trastuzumab+Pertuzumab Group
Drug: Pertuzumab Injection — Pertuzumab injection.
  Arms: Docetaxel+Carboplatin+Trastuzumab+Pertuzumab Group

SUMMARY:
This study is a multicenter, randomized, open-label, parallel Phase III clinical trial. 650 early-stage or locally advanced breast cancer participants will be enrolled and randomly assigned to SHR-A1811 monotherapy group (trial group) or TCbHP treatment group (control group) at a 1:1 ratio. Participants will receive neoadjuvant treatments of SHR-A1811 or TCbHP, while those who have completed neoadjuvant therapy and are suitable for surgery must undergo surgical treatment. The participants will be evaluated on tumor efficacy through postoperative pathological assessment by IRC and pathologists from the research center. The primary endpoint will be tpCR evaluated by IRC. Participants who complete surgical treatment will be followed up for at least 3 years at study endpoints such as EFS, DFS, and DDFS.

ELIGIBILITY:
Inclusion Criteria:

1. Females treated for the first time, 18-75 years old;
2. ECOG score 0-1;
3. Has pathological diagnosis that meets the criteria: confirmed HER2 positive;
4. Results of laboratory tests meet the enrollment requirements;
5. Pregnancy test result must be negative and must agree to contraception;
6. Has signed the informed consent form.

Exclusion Criteria:

1. Confirmed HER2 negative;
2. Has tumor-related medical history or treatment history;
3. Has severe combined disease/medical history and treatment history;
4. Has received treatment with systemic immunostimulants or immunosuppressants;
5. Be allergic to the test drug;
6. Participate in other clinical trials simultaneously;
7. Has received vaccine within 30 days before the first dose;
8. Has received allograft bone marrow transplantation;
9. Has given birth within one year or is breastfeeding;
10. Has history of psychological drug abuse, alcoholism or drug use.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 740 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative total pathologic complete response (tpCR) evaluated by Independent Review Committee (IRC) after finishing neoadjuvant treatments. | From the enrollment of the first subject to the end of the study, it lasted about 36 months.

SECONDARY OUTCOMES:
Postoperative total pathologic complete response (tpCR) evaluated pathologists at the research center after finishing neoadjuvant treatments. | From the enrollment of the first subject to the end of the study, it lasted about 36 months.
Event-free survival (EFS). | Followed up for at least 3 years.
Disease-free survival (DFS). | Followed up for at least 3 years.
Distant disease-free survival (DDFS). | Followed up for at least 3 years.
Objective response rate (ORR) assessed according to the preoperative evaluation utilizing RECIST v1.1 after finishing neoadjuvant treatments. | Followed up for at least 3 years.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shengjing Hospital, China Medical University, Shenyang, Liaoning
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided